CLINICAL TRIAL: NCT03575559
Title: What Friends Are for: Comparing the Effectiveness of an Individual Planning Intervention With Collaborative Planning
Brief Title: TWOgether - From Sport Zero to Sport Hero
Acronym: TWOgether
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); SWPS University of Social Sciences and Humanities (Other); University of Southern Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 100019_169781/1
Record Dates: First submitted 2018-06-18; First posted 2018-07-02 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Physical Activity; Adolescent Behavior; Health Behavior
MeSH Terms: conditions — Motor Activity; Adolescent Behavior; Health Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: Friendship dyads are assigned to the 4 conditions without being informed that 4 conditions exist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individual planning (Experimental): An education and general motivational treatment is provided to each participant. Afterwards, participants are filling in the planning forms, referring to their individual physical activity. Both members of the dyad form up to three own individual plans. They are not allowed to speak to each other. The following behavior change techniques (BCT) are included in the planning intervention protocol: action planning, barrier identification, problem solving (coping planning). Interventions: Behavioral: Individual planning. Behavioral: Education and motivation. Active Comparator: No planning intervention, individual distraction task.
  Interventions: Behavioral: Individual planning; Behavioral: Education and motivation treatment
- Collaborative planning (Experimental): An education and general motivational treatment is provided to each participant. Afterwards, participants are filling in the planning forms together, referring to their joint physical activity. The friendship dyad forms up to three joint plans about engaging in PA together. The following behavior change techniques (BCT) are included in the planning intervention protocol: action planning, barrier identification, problem solving (coping planning). Interventions: Behavioral: Collaborative planning. Behavioral: Education and motivation. Active Comparator: No planning intervention, collaborative distraction task.
  Interventions: Behavioral: Collaborative planning; Behavioral: Education and motivation treatment
- Individual distraction task (Active Comparator): An education and general motivational treatment is provided to each participant. Afterwards, participants have to interpret a short video showing scenes of two different superhero movies. Several questions will be asked about characteristics of the two super heroes in the movie and whether these heroes are comparable. Each participant watches the movie alone and answers all questions by him/herself. Both members of the dyad are not allowed to speak to each other.
  Interventions: Behavioral: Education and motivation treatment
- Collaborative distraction task (Active Comparator): An education and general motivational treatment is provided to each participant. Afterwards, participants have to interpret a short video showing scenes of two different superhero movies together. Several questions ask about the characteristics of the two super heroes in the movie and whether these heroes are comparable. Both members of the dyad watch the movie together and answer the questions conjointly.
  Interventions: Behavioral: Education and motivation treatment

INTERVENTIONS:
Behavioral: Individual planning — Each participant forms up to three action and up to three coping plans individually, without consulting the participating friend, but discussing the plans with the experimenter. CONTENT: The planning materials and forms have the following sections: (a) information on the importance of planning (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans based on the if-then structure. Action plans (referring to when, when, and how the individual will act) as well as coping plans (referring to how to overcome potential difficulties, risky situations or temptations to not engage in physical activity).
  Arms: Individual planning
Behavioral: Collaborative planning — Both friends together create up to three if-then plans on when, where, and how both will implement PA together. In addition, up to three coping plans will be formed together. This jointly developed plan is discussed with the experimenter. CONTENT: The planning materials and forms have the following sections: (a) information on the importance of planning (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans based on the if-then structure. Action plans refers to when, when, and how the individual will act) as well as coping plans (referring to how to overcome potential difficulties, risky situations or temptations to not engage in PA). All materials are formulated using the plural.
  Arms: Collaborative planning
Behavioral: Education and motivation treatment — Adolescents will watch a movie from the Federal Office of Public Health Switzerland including the guidelines of physical activity (PA) for adolescents. All adolescents respond to a quiz afterwards. After the quiz, the experimenter repeats the guidelines for PA based on a brochure that all adolescents can take home with them. In addition, the experimenter asks for barriers and benefits of PA the adolescents perceive. Next to it, the experimenter explains that a weight gain might be possible due to PA in the beginning. Furthermore, the experimenter presents how the data of the accelerometer should look like if one is sufficiently physical active. As a last part self-efficacy as an important aspect of goal success is mentioned. The materials exclude any planning statements.

SUMMARY:
BACKGROUND: The physiological and psychological benefits of regular physical activity (PA) and reduced sedentary behavior are well documented. Nevertheless, the majority of adolescents in western countries, e.g., Switzerland, do not meet the recommendations for moderate to vigorous PA of at least one hour per day. Planning interventions, defined as the creation of plans when, where and how to engage in a behavior change, have been proposed as an effective way of translating intentions into action. AIM: The project aims at closing the empirical gap of the question whether or not planning interventions of PA in adolescents are successful and which planning intervention is the most effective one.

In detail, it is aimed for to examine changes in (daily) moderate to vigorous physical activity in adolescents' friendship dyads following (a) an individual planning intervention, (b) a collaborative planning intervention or (c) one of the two no-planning control conditions. Changes in (daily) physical activity will be examined over a period of 6-months. By investigating the intervention effect systematically by means of daily diaries, long-term follow-ups and objective measurements this project will provide a novel knowledge about individual self-regulating mechanism and social exchange processes as the mediating mechanism of the effectiveness of individual and collaborative planning for health behavior change in adolescents. DESIGN: Single-blind four-arm parallel-group cluster-randomized controlled trial with longitudinal design. The assessment of the main and secondary outcomes is conducted at the baseline, at 1 week after the first intervention session, and at 1-, and 6-month follow-ups. The intervention consists of one planning session and one booster session after 1-month. PARTICIPANTS: The sample will consist of 400 friendship dyads between 14 and 18 years of age. A cluster-randomization will assign participants to one of the two planning groups (collaborative or individual) or one of the two control groups. Both partners of the friendship dyad will complete all questionnaires. OUTCOMES: Physical activity constitutes the main outcome, whereas self-regulatory strategies like planning, self-efficacy, as well as social exchange processes like social support are secondary outcomes.

DETAILED DESCRIPTION:
The physiological and psychological benefits of regular physical activity (PA) and reduced sedentary behavior are well documented. Nevertheless, the majority of adolescents in western countries, e.g., Switzerland, do not meet the recommendations for moderate to vigorous PA of at least one hour per day. However, changing PA seems to be a major challenge even for individuals with good intentions to do so. This phenomenon is the so called intention-behavior gap. Planning interventions have been proposed as an effective way of translating intentions into action. Planning includes action planning (i.e., individual creation of plans when, where and how to engage in a behavior change) and coping planning (i.e., what an individual will do in case barriers arise). So far, good evidence has been found for individual planning increasing PA among adults. Such research with adolescents, however, is in its early stages. Moreover, recent research suggests that an individual's behavior change is also dependent on members of the social network. Consequently, the idea of conjoint planning was introduced recently. Conjoint planning comprises two planning formats, namely collaborative and dyadic planning. Dyadic planning implies creating plans together with a partner, but executing the behavior individually. In contrast, collaborative planning is defined as conjoint planning of at least two individuals when, where and how to perform a behavior together. An example would be "If we go shopping, we will take the bicycles to get there". It is assumed that conjoint planning stimulates social exchange processes between the planning partners. Social exchange processes are interactions between individuals that influence an individual's behavior, emotions, and cognitions and have been shown to play a significant role for health behavior change. A central component of social exchange processes is social support. Regarding PA in adolescents, the influence of peers and friends become increasingly important due to increased autonomy in adolescence. However, past research on health behavior change in adolescents has not yet examined effects of conjoint planning to enhance PA in adolescents. Although a few studies showed promising effects of conjoint planning in adults and adolescents, some important questions still remain open, which will be addressed in this project focusing on individual and collaborative planning. Our research questions and hypotheses are the following:

Research question 1: Is planning an effective strategy to promote PA in adolescents when using daily based measures of PA and long-term follow-ups?

Hypothesis 1.1. Adolescents, who take part in one of the two planning interventions, will show higher levels of (self-reported/objectively measured) PA compared to the control groups when comparing PA on a daily basis, one week (directly after the intervention), one month (after the booster session) and six months after the intervention.

Hypothesis 1.2. Adolescents in the individual and collaborative planning intervention will report higher PA one month and six months after the intervention compared to the control groups.

Research question 2: Do collaborative and individual planning differ regarding their effectiveness to promote PA in adolescents?

Hypothesis 2.1. Adolescents, who take part in the collaborative planning intervention, will show higher levels of (self-reported/objectively measured) PA compared to the individual planning intervention when comparing PA on a daily basis, one week (directly after the intervention), one month (after the booster session) and six months after the intervention.

Hypothesis 2.2. Adolescents in the collaborative planning intervention will report higher PA one month and six months after the intervention compared to the individual planning intervention and the control groups.

Research question 3: Does the planning intervention increase individual self-regulatory processes over time?

Hypothesis 3.1. Adolescents in the individual and collaborative planning intervention will report higher daily self-efficacy one week (directly after the intervention), one month (after the booster session) and six months after the intervention compared to the control groups.

Hypothesis 3.2. Adolescents in the individual and collaborative planning intervention will report higher self-efficacy one month and six months after the intervention compared to the control groups.

Hypothesis 3.3. Adolescents in the individual and collaborative planning intervention will report higher daily (self-reported) planning one week (directly after the intervention), one month (after the booster session) and six months after the intervention compared to the control groups.

Hypothesis 3.4. Adolescents in the individual and collaborative planning intervention will report higher (self-reported) planning one month and six months after the intervention compared to the control groups.

Research question 4: Does the collaborative planning intervention increase social exchange processes over time?

Hypothesis 4.1. Adolescents in the collaborative planning intervention will report higher daily levels of social support one week (directly after the intervention), one month (after the booster session) and six months after the intervention compared to the individual planning condition and the control groups.

Hypothesis 4.2. Adolescents in the collaborative planning intervention will report higher levels of social support one month and six months after the intervention compared to the individual planning condition and the control groups.

Research question 5: What are the underlying mechanisms of the planning interventions in adolescents regarding PA?

Hypothesis 5.1. The effect of the individual planning intervention on daily (self-reported/objectively measured) PA, one week (directly after the intervention), one month (after the booster session) and six months later is mediated by changes in daily individual self-regulatory strategies like self-efficacy, and self-reported planning.

Hypothesis 5.2. The effect of the individual planning intervention on (self-reported) PA, one month and six months later is mediated by changes in individual self-regulatory strategies like self-efficacy, and self-reported planning.

Hypothesis 5.3. The effect of the collaborative planning intervention on daily (self-reported/objectively measured) PA, one week (directly after the intervention), one month (after the booster session) and six months later is mediated by changes in daily levels of social support, as well as by changes in daily individual self-regulatory strategies like self-efficacy, and self-reported planning.

Hypothesis 5.4. The effect of the collaborative planning intervention on (self-reported) PA, one month and six months later is mediated by changes in levels of social support and changes in individual self-regulatory strategies like self-efficacy, and self-reported planning.

Design: This study is designed as a single-blind four-arm parallel-group cluster randomized controlled trial with longitudinal design. The design will comprise a baseline assessment, the intervention and two follow-ups one and six months after baseline. The sample will consist of 400 friendship dyads between 14 and 18 years of age. Recruitment will take place at schools. Therefore, a cluster randomization based upon the schools of all dyads to the four intervention arms is used. In addition, a blocked randomization is used to ensure an equal allocation ration of all a school types (level A; secondary school; vocational school) to the study conditions. All participants being interested in the study, fill in a pre-screening online questionnaire (runin) with the inclusion and exclusion criteria. Afterwards, the friendship dyad will be contacted to make an appointment for the first baseline measurement (T1). Subsequently, adolescents fill in the end-of day diaries and wear the accelerometers for eight days. After this week, the dyads will be invited for the intervention session (T2). All participants will receive an education and general motivational treatment to enhance daily physical activity and are then blocked randomly assigned to one of four intervention conditions: (a) a collaborative planning intervention, in which both adolescents form action and coping plans together to increase daily physical activity together, or (b) an individual planning intervention, in which both adolescents form such action and coping plans individually, or (c) a no-planning control condition, in which both adolescents perform a distraction task together, or (d) a no-planning control condition, in which both adolescents perform a distraction task alone, separately from each other. After the intervention session all adolescents fill in the end-of day diaries and wear the accelerometers for the following seven days. Adolescents of the two planning conditions will receive weekly messages to rethink and adapt their plans with the request to send them to the experimenters. One month (T3) after the intervention all participants are invited for the booster session. Adolescents of the two planning conditions will work on their plans again to adapt or improve them. After this session all participants fill in the end-of day diaries and wear the accelerometers for the following seven days. On a monthly basis all participants of the planning conditions will receive messages to rethink and adapt their plans with the request to send them to the experimenters. Six month after the intervention the participants will be invited to the six-month follow-up (T4). Again, all participants subsequently fill in the end-of day diaries and wear the accelerometers for the following seven days. During all sessions and the daily diaries both partners of the friendship dyad will complete all questionnaires. Self-reports of PA and sedentary behavior, as well as objectively measured PA as the main constructs will be assessed at all time points. Self-regulation constructs (e.g., self-efficacy) will be assessed at time point 1, 3, and 4, whereas social support will be assessed at time T2-T4. In addition, the body weight, height, and body fat tissue will be measured objectively at T1, T3, and T4. The Ethics Committee of the Faculty of Arts and Social Sciences of the University of Zurich, ref: 2017.10.3 approved the study.

Results of this project aims at closing the empirical gap of the question whether planning interventions of PA in adolescents are successful and which planning intervention is the most effective one. By investigating this systematically by means of daily diaries, long-term follow-ups and objective measurements this study will provide novel knowledge about social exchange processes as the mediating mechanism of the effectiveness of collaborative planning for health behavior change in adolescents. Consequently, effective theory-based and evidence-based interventions to promote PA in adolescents can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents (age 14-18)
* Same sex of the adolescents of each friendship dyad
* Access to internet (smartphone or at home)
* Adolescents less active than 1 hour of moderate to vigorous physically active per day
* Adolescents with the intention to be more physically active
* Parental consent at the baseline for adolescents under the age of 16
* Adolescents consent at the baseline

Exclusion Criteria:

* Restrictions on being physically active as assessed by a risk-check form modelled after the Physical Activity Readiness Questionnaire
* Romantic relationship with participating friend
* A BMI below 17
* Insufficient comprehension of the German language
* Pregnancy
* Participating in other intervention programmes targeting physical activity

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective measurement of physical activity | 4 daily diary phases of one week each over a period of 6 month
  Physical activity will be assessed by an accelerometer device ActiGraph (model wGT3X-BT). At each assessment, accelerometer devices will be worn for 7 days (8 days for the first assessment). Accelerometers will be worn by both members of the dyad.
Subjective measurement of daily physical activity | 4 daily diary phases of one week each over a period of 6 month
  Self-reported daily physical activity of all participants is assessed including detailed information on time spent on physical activities, the intensity of each PA and how long each activity has been done together with the friend.
Subjective measurement of physical activity during the past 7 days | Time point one (T1, Month 1) to Time point four (T4; 6 month follow-up)
  Self-reported physical activity of all participants is assessed including detailed information on time spent on physical activities during the past 7 days, the intensity of each PA and how long each activity has been done together with the friend.

SECONDARY OUTCOMES:
Subjective measurement of daily self-efficacy | 4 daily diary phases of one week each over a period of 6 month
  Self-reported daily self-efficacy will be assessed in all adolescents.
Subjective measurement of daily planning | 4 daily diary phases of one week each over a period of 6 month
  Self-reported daily planning of physical activity will be assessed for all adolescents.
Subjective measurement of self-efficacy | Time point one (T1, Month 1) to Time point four (T4; 6 month follow-up)
  Self-reported self-efficacy will be assessed in all adolescents.
Subjective measurement of planning | Time point one (T1, Month 1) to Time point four (T4; 6 month follow-up)
  Self-reported planning of physical activity will be assessed for all adolescents.

OTHER OUTCOMES:
Body mass index | Time point one (T1, Month 1) to Time point four (T4; 6 month follow-up)
  Body mass index (BMI). Certified and standardized body weight scales (OMRON BF 214; measurement error < 5%) and measuring rods will be used. BMI will be calculated as body weight (in kilograms) divided by a square height (in meters).

CONTACTS AND LOCATIONS:
Overall Officials: Theda Radtke, PhD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
In line with the recommendations of the Swiss National Science Foundation the data underlying publications will be shared (anonymised) to make the published results reproducible.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol will be published before the end of the study. In line with the recommendations of the Swiss National Science Foundation the data underlying publications will be shared to make the published results reproducible after submission of the papers.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Derived] Radtke T, Luszczynska A, Schenkel K, Biddle S, Scholz U. A cluster randomized controlled trial comparing the effectiveness of an individual planning intervention with collaborative planning in adolescent friendship dyads to enhance physical activity (TWOgether). BMC Public Health. 2018 Jul 24;18(1):911. doi: 10.1186/s12889-018-5818-6. PMID 30041603
- See also: Information about physical activity — https://www.youtube.com/watch?v=ll9m0sx9uAI